CLINICAL TRIAL: NCT05321303
Title: The Effect of Serious Game Developed for Nursing Education on Students' Knowledge Level, Critical Thinking and Problem Solving Skills
Brief Title: The Effect of Serious Game Developed for Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Afra CALIK, Research Asisstant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21/06-26
Record Dates: First submitted 2022-02-23; First posted 2022-04-11 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Education, Nursing; Critical Thinking; Problem Solving; Self-Confidence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Serious game Experimental group (Experimental): The participants spend on one "MetaHospital" scenario in which Nursing Care (management of diabetic ketoacidosis).
  Interventions: Other: Serious Game
- Experimental: Standardized Patients Control group (Experimental): The participants spend one scenario 10 minutes; on a scenario designed to train Nursing Care (management of diabetic ketoacidosis).
  Interventions: Other: Standard Patients

INTERVENTIONS:
Other: Serious Game — Each participant of the Serious game group played 1 scenario of "MetaHospital", a screen-based simulation on the management of diabetic ketoacidosis. Immediately after the serious game was played, 5 open-ended questionnaires were sent to the students to evaluate the game usability.
  Arms: Experimental: Serious game Experimental group
Other: Standard Patients — Each participant of the standardized patient's group played 1 scenario on the management of diabetic ketoacidosis and then a 30-minute analysis session with the trainer joined.
  Arms: Experimental: Standardized Patients Control group

SUMMARY:
The aim of the study is to assess whether students' knowledge level, critical thinking, and problem-solving skills have increased after the serious game and standard patients practice.

DETAILED DESCRIPTION:
This study aims to answer the following problematic: How to improve the learning of satisfaction and self-confidence, knowledge Levels, problem-solving, critical thinking skills in serious game, and standardized patients practice for students. This study tests nursing care skills learning in a serious game on diabetic ketoacidosis management designed scenarios.

50 students in nursing in 2nd year will participate in the experiment. They will be randomized into 2 groups:

Standardized patient Control group (25 participants): The participants spend one scenario 10 minutes; a scenario designed to train Nursing Care (management of diabetic ketoacidosis).

Serious game Experimental group (25 participants): The participants spend on one "MetaHospital" scenario in which Nursing Care (management of diabetic ketoacidosis).

Before the serious game and standard patients practice, students will be asked to fill out a questionnaire on their knowledge level, satisfaction and self-confidence, critical thinking, and problem-solving skills in line with the purpose of the study. The form was submitted to evaluate the usability of the game immediately after the students played the serious game.

Students will be given an information session regarding the case prior to the standard patient practice. Following that, each student will do a standard patient practice for 10 minutes once. After 25 students have finished the application, a 30-minute analysis session with the trainer will be placed. The knowledge levels, satisfaction and self-confidence, critical thinking, and problem-solving skills questionnaires will be filled out again after the session.

Before the serious game application, and after the students have been notified about the game, each student will be provided a username and password for the game login. For one day, students will have unrestricted access to the game. All students participating in the activities will be asked to complete a questionnaire about their knowledge level, satisfaction and self-confidence, critical thinking, and problem-solving abilities.

After the two applications are finished, a questionnaire regarding students' interests, knowledge level, satisfaction and self-confidence, critical thinking, and problem-solving skills will be provided to them one month later to evaluate their learning retention. Finally, the researcher will conduct focus group interviews with students to hear about their experiences.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students who have taken the Internal Medicine Nursing course
* Students willing and willing to participate in the research

Exclusion Criteria:

* Students who are absent from the Internal Medicine Nursing course
* Students who did not agree to participate in the study
* Students experiencing standard patient practice

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Knowledge Levels Questionnaire | Five weeks
  In order to determine the knowledge level of the students about the diabetic ketoacidosis case, the opinions of 3 experts (diabetes nurse, academician working in the field of diabetes) were taken, prepared by the researcher. There are 10 questions in total and each question is 1 point.
Student Satisfaction and Self-Confidence in Learning Scale | Five weeks
  The scale consists of two sub-dimensions (satisfaction with learning and self-confidence) in five-point Likert type. The total number of items is 13. The minimum score obtained from the scale is 17, the highest score is 61.
Critical Thinking Disposition Scale | Five weeks
  The scale consists of 49 items and 5 subscales (metacognition, flexibility, systematicity, perseverance-patience, open-mindedness). The range of points that can be obtained from the scale varies between 49-245. An increase in the score indicates that critical thinking also increases.
Problem Solving Inventory | Five weeks
  It is a Likert-type scale consisting of 35 items and scored between 1-6. As the score obtained from the scale increases, problem solving skills decrease. The lowest score that can be obtained from the scale is 32, and the highest score is 192.

SECONDARY OUTCOMES:
Student experience: Qualitative Interviewing | up to four weeks
  40-50 minutes of focus group discussions will be held with students in order to better determine the effectiveness of the methods used, to share experiences and to support future studies.
Serious Game Experience: | up to one day
  It is a data form consisting of 6 open-ended questions to evaluate the game usability immediately after playing the serious game.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF